CLINICAL TRIAL: NCT01563588
Title: Post Therapeutic Support and Rehabilitation Protocol in Hydrothermal Centers for Breast Cancer Patients in Complete Remission: a Multicenter Prospective Randomized Trial Testing the Intervention Versus Best Supportive Care
Brief Title: Support and Rehabilitation Protocol for Non Metastatic Breast Cancer Patients in Complete Remission After Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment lasted longer than expected and expected number of patients could not be matched in time.
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Principal Investigator, Philippe Chollet, Professor Yves-Jean Bignon, Centre Jean Perrin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACThe; 2008-A 01606 - 49 (Registry Identifier: AFSSAPS (France))
Record Dates: First submitted 2012-02-22; First posted 2012-03-27 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Non Metastatic Breast Cancer
Keywords: breast cancer; chemotherapy; first line treatment; treatments include a chemotherapy; last treatment not performed more than 9 months earlier
MeSH Terms: conditions — Breast Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dietary and physical training (Experimental): 12 days session of physical training, dietary education, physiotherapy and SPA cares in small group (less than 12 women) delivered in hydrothermal centers
  Interventions: Behavioral: dietaty education, physical training, physiotherapy and SPA cares
- control (No Intervention): dietary counseling by a dietetician in the anticancer hospital

INTERVENTIONS:
Behavioral: dietaty education, physical training, physiotherapy and SPA cares — 12 days session of daily physical training, dietary education, physiotherapy and SPA cares in small group (less than 12 women) delivered in hydrothermal centers
  Arms: dietary and physical training

SUMMARY:
Many breast cancer patients (BCP) will gain weight during chemotherapy and about 10% of them are able to find back to their initial weight after all treatments are finished. Other studies have shown that overweight at diagnosis was associated to a twice higher risk of relapse while a weight gain during treatments increased by 30% to 50% the risk of relapse. In western countries, 75% of BCP have insufficient physical activity. Dietary and activity programs seem to be able to significantly reduce the mortality risk after breast cancer.

The investigators performed a prospective randomized trial consisting in dietary counseling, physical training and physiotherapy in hydrothermal centers. Intervention were delivered in small group session lasting 12 days. SPA cares were offered to patients. Patients in the control group also received dietary counseling given by a dietetician inside anticancer hospital, and were asked to perform more physical activities. Main endpoints of the trial addressed quality of life (SF36) one year after inclusion, weight reduction, anxiety/depression (HAD), sleep quality and long term compliance to instructions. An economic study was associated to the protocol, for volunteers only.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* treatment including a chemotherapy
* in complete remission
* last treatment in the last 9 months before inclusion
* signed consent

Exclusion Criteria:

* metastatic disease
* relapse
* women enable to have physical activity
* heart disease or any pathology preventing physical activity

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quality of life (SF36) | one year after inclusion
  Quality of life was measured with the SF36 questionnaire before randomization, at 6, 12, 18, 24 and 36 months. The difference at one year was the main endpoint.

SECONDARY OUTCOMES:
Anxiety/depression scores (HAD) | inclusion, 6, 12, 18, 24, 36 months
  HAD questionnaire is a validated instrument that complete the SF36 QoL questionnaire.
Weight and morphometric measures | inclusion, 6, 12, 18, 24, 36 months
  Weight(kg), impedancemetry, hip/waist circumference are needed to characterize eventual weight changes in both allocation groups
Sleep quality | inclusion, 6, 12, 18, 24, 36 months
  6 questions are asked: it rates the delay before sleep onset, the lenght of sleep, the number of awakening, the lenght of wake periods during the night, the concentration/alertness after sleep, and the fatigue in the morning.
economic figures | during 2 years after inclusion
  health related costs, health insurance costs, social costs

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Jean Perrin, Clermont-Ferrand, Puy de Dome
  - Pole Santé-République, Clermont-Ferrand, Puy de Dome

REFERENCES:
- See also: URL to Centre Jean Perrin main page — http://www.cjp.fr/